CLINICAL TRIAL: NCT00453570
Title: Immunogenicity and Safety of Pentaxim as 3 Doses Primary Vaccination Followed by a Booster Dose at 18 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E2I42
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Diphtheria; Tetanus; Haemophilus Influenzae Type b; Pertussis; Poliomyelitis
Keywords: Diphteria; Tetanus; Haemophilus influenzae type b; Poliomyelitis; Pertussis
MeSH Terms: conditions — Diphtheria; Tetanus; Haemophilus Infections; Whooping Cough; Poliomyelitis | interventions — Tetanus Toxoid; Pentavac; Hiberix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): DTacP IPV// PRP~T combined vaccine at 2, 3 and 4 months of age, and a booster dose at 18-20 months of age.
  Interventions: Biological: Diphtheria, Tetanus, Polio, Acellular Pertussis and Hib
- 2 (Experimental): DTacP-IPV// PRP~T combined vaccine at 3, 4 and 5 months of age and a booster dose at 18-20 months of age.
  Interventions: Biological: Diphtheria, Tetanus, Polio, Acellular Pertussis and Hib
- 3 (Active Comparator): Control vaccines at 3, 4 and 5 months of age and a booster dose at 18-20 months of age
  Interventions: Biological: Diphtheria, Tetanus, & Acellular Pertussis Combined, Absorbed

INTERVENTIONS:
Biological: Diphtheria, Tetanus, Polio, Acellular Pertussis and Hib — 0.5 mL, IM
  Other Names: PENTAXIM™
  Arms: 1
Biological: Diphtheria, Tetanus, Polio, Acellular Pertussis and Hib — 0.5 mL, IM
  Other Names: PENTAXIM™
  Arms: 2
Biological: Diphtheria, Tetanus, & Acellular Pertussis Combined, Absorbed — 0.5 mL, IM
  Other Names: DTacP, Act-HIB™ and IMOVAX Polio™
  Arms: 3

SUMMARY:
As per request by the Heath Authorities, the present clinical study will assess the immunogenicity and safety of sanofi pasteur's DTacP-IPV// PRP~T combined vaccine (PENTAXIM™) as a three-dose primary vaccination at 2, 3, and 4 months of age or 3, 4 and 5 months of age followed by a booster dose at 18-20 months of age as compared to commercially available DTacP, Hib conjugate (Act-HIB™) and IPV (IMOVAX Polio™) monovalent vaccines in order to meet the requirements for registration of the product in People's Republic of China.

ELIGIBILITY:
Inclusion Criteria :

* Aged 2 months (60 to 74 days) inclusive on the day of inclusion
* Born at full term pregnancy (³36 weeks) with a birth weight ≥ 2.5 kg
* Informed consent form signed by the parent(s) or other legal representative
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria :

* Participation in another clinical trial in the 4 weeks preceding the trial inclusion
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received in the past
* Any vaccination performed or planned in the 4 weeks preceding the first trial visit (except BCG and Hepatitis B, which can not be given within 8 days before the first study visit)
* Vaccination planned in the 4 weeks following any trial vaccination (except BCG and Hepatitis B, which can not be given within 8 days before or after the study vaccine(s) administration)
* History of diphtheria, tetanus, pertussis, poliomyelitis, Haemophilus influenzae type b infection (confirmed either clinically, serologically or microbiologically)
* Clinical or serological evidence of systemic illness including Hepatitis B, Hepatitis C and/or HIV infection
* Previous vaccination against the diphtheria, tetanus, pertussis, poliomyelitis diseases or Haemophilus influenzae type b infection with the trial vaccine or another vaccine
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of/current seizures
* Febrile illness (axillary temperature ≥ 37.1°C) or acute illness on the day of inclusion

Ages: 60 Days to 74 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 792 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of DTacP-IPV//PRP~T combined vaccine | 1 Month post-dose 3

SECONDARY OUTCOMES:
To provide information concerning the safety of DTacP-IPV//PRP~T combined vaccine | 19 months post-dose 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Nanning, Guangxi, China

REFERENCES:
- [Derived] Li RC, Li FX, Li YP, Hou QM, Li CG, Li YN, Chen FS, Hu XZ, Su WB, Zhang SM, Fang HH, Ye Q, Zeng TD, Liu TX, Li XB, Huang YN, Deng ML, Zhang YP, Ortiz E. Antibody persistence at 18-20 months of age and safety and immunogenicity of a booster dose of a combined DTaP-IPV//PRP approximately T vaccine compared to separate vaccines (DTaP, PRP approximately T and IPV) following primary vaccination of healthy infants in the People's Republic of China. Vaccine. 2011 Nov 21;29(50):9337-44. doi: 10.1016/j.vaccine.2011.09.131. Epub 2011 Oct 14. PMID 22001281
- [Derived] Li RC, Li FX, Li YP, Hou QM, Li CG, Li YN, Chen FS, Hu XZ, Su WB, Zhang SM, Fang HH, Ye Q, Zeng TD, Liu TX, Li XB, Huang YN, Deng ML, Zhang YP, Ortiz E. Immunogenicity and safety of a pentavalent acellular pertussis combined vaccine including diphtheria, tetanus, inactivated poliovirus and conjugated Haemophilus Influenzae type b polysaccharide for primary vaccination at 2, 3, 4 or 3, 4, 5 months of age in infants in China. Vaccine. 2011 Feb 24;29(10):1913-20. doi: 10.1016/j.vaccine.2010.12.103. Epub 2011 Jan 8. PMID 21219984
- See also: Related Info — http://www.sanofipasteur.com